CLINICAL TRIAL: NCT07321132
Title: The Effect of Yoga on the Level of Burnout and Happiness in Midwifery Students: Randomized Controlled Study
Brief Title: Effects of Yoga on Burnout and Happiness in Midwifery Students
Acronym: EYBHMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Ayşe ÇATALOLUK, Ass. Prof. Dr., Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TOGUE-13232362-804.01-295714
Record Dates: First submitted 2025-12-02; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Midwifery Students
Keywords: yoga; health; midwifery students; burnout; happiness; well-being
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: The research was conducted as a randomized controlled experimental study. Participants were devided into two groups: yoga exercise group and control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Practice Program (Experimental): Yoga Practice (Weeks 1-6): Each yoga session began with a 5-minute breathing exercise, which formed the first phase of the practice. This segment included a combination of different breathing techniques. Students were guided to breathe slowly and rhythmically while listening to calming background music, helping them first become aware of their natural breath and then regulate it consciously. Each session started with three selected breathing techniques, such as yogic breathing, alternate nostril breathing (nadi shodhana), and the 4-7-8 breathing method. Following the breathing exercises, participants engaged in a 40-minute asana (posture) practice, which included five standing poses, two transitional poses, and five seated poses, or the reverse order, depending on the session structure. Each yoga session concluded with 5 to 10 minutes of relaxation and meditation, promoting physical and mental calmness.
  Interventions: Other: Yoga Practice (Non-pharmacological, Non-device)
- Control group (No Intervention): After randomization, students assigned to the control group were informed about the study. Written and verbal informed consent was obtained, and the socio-demographic information form was completed. No intervention was applied to the students in this group. They were only asked to complete the data collection forms (MBI-SS and OHQ-SF).

INTERVENTIONS:
Other: Yoga Practice (Non-pharmacological, Non-device) — Each yoga session began with a 5-minute breathing exercise, which formed the first phase of the practice. This segment included a combination of different breathing techniques. Students were guided to breathe slowly and rhythmically while listening to calming background music, helping them first become aware of their natural breath and then regulate it consciously. Each session started with three selected breathing techniques, such as yogic breathing, alternate nostril breathing (nadi shodhana), and the 4-7-8 breathing method. Following the breathing exercises, participants engaged in a 40-minute asana (posture) practice, which included five standing poses, two transitional poses, and five seated poses, or the reverse order, depending on the session structure. Each yoga session concluded with 5 to 10 minutes of relaxation and meditation, promoting physical and mental calmness.
  No drugs, medical devices, or invasive procedures were used during the intervention.
  Arms: Yoga Practice Program

SUMMARY:
The health sector constitutes a highly stressful environment not only for professionals working in the field but also for students undergoing training. In particular, students studying in the health sciences experience stress due to various factors such as intensive theoretical coursework, practical training, clinical responsibilities, and shift duties. For midwifery students, who receive education in areas requiring a high level of responsibility such as women's health, the childbirth process, and newborn care, this level of stress may be even greater. Prolonged and intense stress can lead to the development of burnout among students, which may negatively affect psychological well-being, happiness, and academic performance.

In recent years, mindfulness-based practices have gained prominence as effective approaches for coping with stress, enhancing psychological resilience, and supporting mental well-being. One such practice is yoga, which is a holistic approach that includes physical postures, breathing exercises, relaxation techniques, and meditation. Previous studies have demonstrated that yoga practices are effective in reducing stress, anxiety, depression, and burnout, while enhancing happiness, life satisfaction, and self-awareness. These findings indicate that yoga and similar practices are particularly beneficial for students studying in health-related fields.

Accordingly, the present study was conducted using a randomized controlled experimental design to evaluate the effects of yoga practice on burnout and happiness levels among midwifery students. The study was carried out with second-year students enrolled in the Midwifery Department of the Faculty of Health Sciences at Tokat Gaziosmanpaşa University. Students were randomly assigned to either the experimental or control group. The experimental group participated in 60-minute yoga sessions three times per week for six weeks, while no intervention was applied to the control group. Burnout and happiness levels of the students were assessed using the Maslach Burnout Inventory-Student Form and the Oxford Happiness Questionnaire-Short Form. The findings of this study are expected to contribute to the literature by highlighting the importance of interventions that support the mental health of midwifery students.

DETAILED DESCRIPTION:
Mental well-being is of great importance for midwifery students to effectively utilize their professional skills. High school and university life may create stress for students due to structured and compulsory activities aimed at specific goals, such as passing examinations, fulfilling academic responsibilities, and obtaining a diploma. Prolonged exposure to stress may lead to burnout, which manifests as physical, emotional, and mental exhaustion and is considered a consequence of chronic stress.

Happiness is defined as the frequent experience of positive emotions, the relatively infrequent experience of negative emotions, and a high level of life satisfaction. It is associated with the prevalence of positive feelings such as trust, hope, and joy, as well as satisfaction derived from various life domains. Students' academic achievement is influenced by factors such as self-esteem, self-efficacy, motivation, and coping skills for managing stress.

In recent years, mind-body practices such as yoga and meditation have become increasingly widespread in educational institutions to help students cope with stress and enhance cognitive functioning. Yoga is a holistic practice consisting of postures (asana), breathing exercises (pranayama), and meditation, and it has been shown to reduce stress and anxiety while supporting overall well-being and cognitive processes. Studies have demonstrated that yoga practices are particularly effective in reducing perceived stress, enhancing well-being, and fostering positive emotions such as empathy and compassion among students in health-related fields.

In this context, the present study aims to compare burnout and happiness levels among midwifery students by forming experimental and control groups consisting of students who practice yoga and those who do not.

ELIGIBILITY:
Inclusion Criteria:

Female midwifery students. Not exercising at least two days per week. Not practicing yoga or other mindfulness-based activities. Able to attend scheduled yoga sessions at the designated location.

Exclusion Criteria:

Presence of musculoskeletal, neuromuscular, or chronic systemic conditions preventing yoga practice.

Recent surgical procedures. Declined to provide consent for participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Midwifery students for women
Enrollment: 72 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2023-12-16 (Actual); Study Completion 2023-12-16 (Actual)

PRIMARY OUTCOMES:
Maslach Burnout Inventory - Student Scale (MBI-SS) | Post-intervention at Week 6 for experimental group, Baseline (Week 0) for control group
  The scale consists of 13 items and includes three subscales: exhaustion, cynicism, and efficacy. The exhaustion subscale measures chronic fatigue and tension resulting from academic responsibilities. The cynicism subscale measures indifference toward school-related activities and a detached, disengaged attitude toward academic tasks. The efficacy subscale measures students' perception of their own academic competence.
  Score Range: 0-6 per item; higher scores on exhaustion and cynicism indicate worse burnout, while higher scores on efficacy indicate better perceived competence.

SECONDARY OUTCOMES:
Oxford Happiness Questionnaire short form (OHQ-SF) | Post-intervention at Week 6 for experimental group, Baseline (Week 0) for control group
  The scale consists of 7 items and measures overall happiness. Items 1 and 7 are reverse-coded. Response options range from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate higher levels of happiness.
  Score Range: 1-5 per item; higher scores indicate greater happiness.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpaşa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No